CLINICAL TRIAL: NCT03907683
Title: Phase 1 Clinical Trial to Develop a Personalized Adaptive Text Message Intervention Using Control Systems Engineering Tools to Increase Physical Activity in Early Adulthood
Brief Title: Random Assignment of Intervention Messages for Developing Personalized Decision Rules to Promote Physical Activity
Acronym: RandomAIM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, David E Conroy, Professor, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00009455; R01HL142732 (NIH)
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Random Messaging (Experimental): Participants receive 0-5 messages/day from the Random AIM app. Messages are only delivered outside of a participant-specific Do Not Disturb window (e.g., 11pm-8am). Messages are selected randomly from three content domains: Move More (40%), Sit Less (40%), and Inspirational Quotes Unrelated to Movement (20%). Half of the messages are accompanied by images. Message selection and timing are determined randomly each night for the following day.
  Interventions: Behavioral: Short Message with Text and Optional Image

INTERVENTIONS:
Behavioral: Short Message with Text and Optional Image — Messages can be up to 256 characters of text and with or without an image. "Move more" and "sit less" messages were written to target established cognitive and affective constructs associated with physical activity (e.g., prompts to action plan, guidance for maximizing pleasure by regulating intensity).

SUMMARY:
Our goal is to develop personalized decision rules for selecting the frequency, timing, and content of messages to promote physical activity. The objective of this project is to develop personalized dynamical models of physical activity (PA) under different weather and temporal conditions as well as in response to different types of intervention messages. This approach relies on having extensive observations within the person under varying conditions to develop a dynamical model of how different conditions interact with each other to predict how behavior changes in response to text messages. Complementary sub-models will be estimated for each participant to describe their behavioral responses under different weather conditions. Healthy but insufficiently active young adults (n=80) will wear an activity monitor and receive a variety of randomly-timed and randomly-selected notifications via smartphone. GPS coordinates at the time of messages delivery and receipt are recorded and used to look up weather indices at that location at that time. The work is exploratory/descriptive as we will be developing models to describe participants' responses to messages under different weather conditions. This work is needed to develop the decision rules for a subsequent behavioral intervention that will be developed and tested in a future project.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of reading, speaking and understanding English and of giving informed consent.
* Participants between the ages of 18-29 years.
* Participants must be free of visual impairment that would interfere with the use of a smartphone.
* Participants must own and carry an iPhone (running iOS version 10 or higher) or Android (running operating system 7 or higher) smartphone during waking hours.

Exclusion Criteria:

* Participants engaging in 90 or more minutes of moderate- or greater intensity PA each week.
* Participants engaged in organized programs with mandated physical activity (e.g., varsity sports, ROTC).
* Participants with contraindications to normal physical activity on the Physical Activity Readiness Questionnaire.
* Participants who require an assistive device for mobility or have any other condition that may limit or prevent participation in moderate-intensity physical activity.
* Participants who are pregnant or planning to become pregnant within the next 6 months.
* Participants with a prior diagnosis of cancer, cardiovascular disease, diabetes or metabolic syndrome.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Conroy, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hojjatinia S, Hojjatinia S, Lagoa CM, Brunke-Reese D, Conroy DE. Person-specific dose-finding for a digital messaging intervention to promote physical activity. Health Psychol. 2021 Aug;40(8):502-512. doi: 10.1037/hea0001117. PMID 34618498

RESULTS

PARTICIPANT FLOW:
Groups:
- Random Messaging: Participants receive 0-6 messages/day from the Random AIM app. Messages are only delivered outside of a participant-specific Do Not Disturb window (e.g., 11pm-8am). Messages are selected randomly from three content domains: Move More (40%), Sit Less (40%), and Inspirational Quotes Unrelated to Movement (20%). Half of the messages are accompanied by images. Message selection and timing are determined randomly each night for the following day.
  Short Message with Text and Optional Image: Messages can be up to 256 characters of text and with or without an image. "Move more" and "sit less" messages were written to target established cognitive and affective constructs associated with physical activity (e.g., prompts to action plan, guidance for maximizing pleasure by regulating intensity).
Period: Overall Study
Arm/Group | Random Messaging
Started | 82
Completed | 80
Not Completed | 2
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Random Messaging
Number analyzed (Participants) | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 82
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 78
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 19
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 47
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 82

OUTCOME MEASURES:

1. Primary Outcome: Change in Moderate (or Higher) Physical Activity Duration Following Message Receipt
Description: Fitbit-assessed minutes with step counts >= 100 steps/min in 15-minute epochs (steady states represent the change in expected step counts if a message was delivered versus if the message was not delivered)
Time Frame: 15-minute epochs for the remainder of the walking day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Random Messaging
Number analyzed (Participants) | 80
minutes
  Weekday Move More Messages (person-specific steady state estimate) | 0.16 (0.69)
  Weekday Sit Less Messages (person-specific steady state estimate) | 0.13 (0.69)
  Weekday Inspirational Quote Messages (person-specific steady state estimate) | 0.25 (1.23)
  Weekend Move More Messages (person-specific steady state estimate) | 0.31 (1.44)
  Weekend Sit Less Messages (person-specific steady state estimate) | 0.28 (0.95)
  Weekend Inspirational Quote Messages (person-specific steady state estimate) | 0.11 (1.51)
Statistical Analysis 1: Comparison: Random Messaging; Null hypothesis was that the mean steady state response to weekday move more messages would not differ from zero; Test type: Superiority; p = 0.037, t-test, 2 sided; Mean Difference (Final Values) = 0.16412, 95% CI 2-sided [.0098 to 0.3185], Standard Error of Mean .08
Statistical Analysis 2: Comparison: Random Messaging; Null hypothesis was that the mean steady state response to weekday sit less messages would not differ from zero; Test type: Superiority; p = .106, t-test, 2 sided; Mean Difference (Net) = .12538, 95% CI 2-sided [-0.0274 to 0.2781], Standard Error of Mean 0.07674
Statistical Analysis 3: Comparison: Random Messaging; Null hypothesis was that the mean steady state response to weekday inspirational quote messages would not differ from zero; Test type: Superiority; p = .076, t-test, 2 sided; Mean Difference (Net) = .24738, 95% CI 2-sided [-.0262 to .5210], Standard Error of Mean 0.13746
Statistical Analysis 4: Comparison: Random Messaging; Null hypothesis was that the mean steady state response to weekend move more messages would not differ from zero; Test type: Superiority; p = .062, t-test, 2 sided; Mean Difference (Net) = 0.30563, 95% CI 2-sided [-.0156 to .6268], Standard Error of Mean 0.16136
Statistical Analysis 5: Comparison: Random Messaging; Null hypothesis was that the mean steady state response to weekend sit less messages would not differ from zero; Test type: Superiority; p = 0.11, t-test, 2 sided; Mean Difference (Net) = .27700, 95% CI 2-sided [.0645 to .4895], Standard Error of Mean 0.10676
Statistical Analysis 6: Comparison: Random Messaging; Null hypothesis was that the mean steady state response to weekend inspirational quote messages would not differ from zero; Test type: Superiority; p = .523, t-test, 2 sided; Mean Difference (Net) = 0.10837, 95% CI 2-sided [-0.2279 to 0.4447], Standard Error of Mean 0.16895

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Random Messaging
All-Cause Mortality (participants affected / at risk) | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 0/82

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic was declared in March 2020 during enrollment and data collection. Some participants completed data collection before the pandemic; others completed data collection during the pandemic. The pandemic adversely impacted physical activity worldwide and may have impacted results from this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT03907683/Prot_SAP_000.pdf